CLINICAL TRIAL: NCT02408692
Title: Emergency Contraception and Body Weight: Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Medical Research Foundation, Oregon (Other)
Responsible Party: Principal Investigator, Alison Edelman, Associate Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OHSU IRB 11419
Record Dates: First submitted 2015-03-27; First posted 2015-04-03 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Contraception; Body Weight
Keywords: Emergency contraception; Obese BMI; Normal BMI
MeSH Terms: conditions — Body Weight | interventions — Contraception, Postcoital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal BMI ECx1 (Active Comparator): 5 normal weight women (BMI<25 kg/m2) taking 1.5mg LNG
  Interventions: Drug: ECx1
- Obese BMI ECx1 (Active Comparator): 5 obese women (BMI >30 kg/m2) taking 1.5mg LNG
  Interventions: Drug: ECx1
- Obese BMI ECx2 (Active Comparator): 5 obese women (BMI >30 kg/m2) taking 3mg LNG
  Interventions: Drug: ECx2

INTERVENTIONS:
Drug: ECx1 — At the first treatment visit, all women will be given the study drug (1.5 mg of levonorgestrel) and several blood samples will be taken over 2.5 hours). After this visit, women with a BMI of <25 kg/m2 will have completed study participation.
  Other Names: Next choice; Emergency Contraception
  Arms: Normal BMI ECx1; Obese BMI ECx1
Drug: ECx2 — At the first treatment visit, all women will be given the study drug (1.5 mg of levonorgestrel) and several blood samples will be taken over 2.5 hours). For women with a BMI of 30kg/m2 and greater, one additional visit will be required and study drug (3 mg of levonorgestrel) will be given and several blood samples will be taken over 2.5 hours)
  Other Names: Next choice; Emergency Contraception
  Arms: Obese BMI ECx2

SUMMARY:
The purpose of this research study is to determine how body weight changes the drug level of an emergency contraceptive pill containing a hormone called levonorgestrel (LNG). This emergency contraceptive is available to women without a prescription, but has recently been found to not work as well to prevent pregnancies in women of higher body weight. The overall goal of this research is to improve the effectiveness of contraception for women, no matter their weight.

DETAILED DESCRIPTION:
To determine if differences exist in the pharmacokinetics (PK) of levonorgestrel-based emergency contraception (LNG-EC) in obese and normal body mass index (BMI) users and test whether doubling the dose of LNG-EC in obese women increases total and free LNG serum concentrations.

We enrolled healthy, reproductive-age women with obese and normal BMIs received 1.5 mg LNG orally and then in a subsequent menstrual cycle, the obese group also received 3 mg LNG. Total and free LNG PK parameters were obtained via serum samples through an indwelling catheter at 0, 0.5, 1, 1.5, 2, and 2.5 h. The primary outcome was the difference in total and free LNG concentration maximum (Cmax) between ECx1 and ECx2 in the obese group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between the ages of 18 and 35
* Subjects are in good general health
* Subjects have regular menstrual cycles (between 21 and 35 days)
* Subjects are willing to use condoms (if you are sexually active with a male partner), subjects are willing to not have sex with men during the study, or subjects have had a tubal ligation (or have a partner who has had a vasectomy) or subjects have a copper intrauterine device (IUD).

Exclusion Criteria:

* Metabolic disorders including uncontrolled thyroid dysfunction and Polycystic Ovarian Syndrome
* Impaired liver or renal function
* Actively seeking or involved in a weight loss program (must be weight stable)
* Pregnancy, breastfeeding, or seeking pregnancy; recent (8 week) use of hormonal contraception
* Current use of drugs that interfere with metabolism of sex steroids
* Smokers.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
PI acknowledges willingness to share data and materials with other investigators through established means. Data will be presented via presentation and publication. Transfer of resources is subject to the acceptance of a Materials Transfer Agreement as required by policy at OHSU. OHSU complies with NIH policy on Sharing Research Data.

REFERENCES:
- [Result] Edelman AB, Cherala G, Blue SW, Erikson DW, Jensen JT. Impact of obesity on the pharmacokinetics of levonorgestrel-based emergency contraception: single and double dosing. Contraception. 2016 Jul;94(1):52-7. doi: 10.1016/j.contraception.2016.03.006. Epub 2016 Mar 18. PMID 27000996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal BMI ECx1 | Obese BMI ECx1 | Obese BMI ECx2
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal BMI ECx1 | Obese BMI ECx1 | Obese BMI ECx2 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration Between Normal and Obese BMI Women Ingesting 1.5mg Levonorgestrel
Description: Pharmacokinetic sampling at 0, 0.5, 1, 1.5, 2, and 2.5 hours were performed after ingestion of 1.5mg of levonorgestrel
Time Frame: Follicular phase of menstrual cycle and PK sampling at 0, 0.5, 1, 1.5, 2, 2.5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal BMI ECx1 | Obese BMI ECx1 | Obese BMI ECx2
Number analyzed (Participants) | 5 | 5 | 0
ng/mL | 10.3 (2.47) | 5.57 (2.76) |

2. Secondary Outcome: Maximum Serum Concentration Between Obese BMI Women Ingesting 1.5mg of Levonorgestrel and Then the Same Obese BMI Women Ingesting 3mg Levonorgestrel
Description: Pharmacokinetic sampling at 0, 0.5, 1, 1.5, 2, and 2.5 hours were performed after ingestion of 3mg of levonorgestrel
Time Frame: Follicular phase of menstrual cycle
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal BMI ECx1 | Obese BMI ECx1 | Obese BMI ECx2
Number analyzed (Participants) | 0 | 5 | 5
ng/mL |  | 5.57 (2.48) | 10.52 (2.76)

ADVERSE EVENTS:
Time Frame: 30 minutes after study medication dosing.
Arm/Group | Normal BMI ECx1 | Obese BMI ECx1 | Obese BMI ECx2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal BMI ECx1 (N=5) | Obese BMI ECx1 (N=5) | Obese BMI ECx2 (N=5)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes